CLINICAL TRIAL: NCT05446207
Title: Effects Of Relaxing Music Therapy Along With Task-Oriented Training On Balance And Functional Independence In Patients With Chronic Stroke: A Randomized Clinical Trial
Brief Title: Effects of Music Therapy Along With Task-Oriented Training on Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Dr. Ayesha Jamil, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hafsa Zahid
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hemiplegia
Keywords: Stroke, Music Therapy, Task-oriented training, Balance, Functional Independence
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will be single blinded study in which the outcome assessor will be unaware of the treatment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): This group will receive routine physiotherapy with task oriented training. This protocol will be given for 3 alternative days per week. Each session will be of 45 minutes. Data will be collected at baseline, at 4th week and at 8th week.
  Interventions: Other: Routine Physiotherapy and Task-oriented Training
- Group B (Experimental): This group will receive passive music therapy and routine physiotherapy with task oriented training. This protocol will be given for 3 alternative days per week. Each session will be of 60 minutes. Data will be collected at baseline, at 4th week and at 8th week.
  Interventions: Other: Music Therapy and Task oriented Training with Routine Physiotherapy

INTERVENTIONS:
Other: Routine Physiotherapy and Task-oriented Training — The routine physiotherapy treatment will include TENS and Hot pack. The task oriented training for lower extremity will include walking training on the ground, equal weight bearing sit-to-stand exercises, resistance exercises e.g. leg press, leg extension, and leg curl and reaching tasks for improving balance. There will be a rest period of 5 minutes between each set of training.
  Arms: Group A
Other: Music Therapy and Task oriented Training with Routine Physiotherapy — Relaxing Music will be provided through headphones having voice cancellation property for 15 minutes.
  Arms: Group B

SUMMARY:
Previous studies discussed the effects of music therapy and task oriented training on motor functions of stroke separately but no study is found in which effects of both techniques are studied. In this study, we are going to find the effects of task oriented training with or without music therapy.

DETAILED DESCRIPTION:
Stroke is a neurological condition, which can promote disability and increase the susceptibility to secondary complications along the patient's life. Stroke issue incorporates motor dysfunction, Cognition, daily activity and sensory weaknesses. Music Therapy appears to affect physiological phenomena such as blood pressure, heartbeat, respiration, and mydriasis as well as emotional aspects such as mood and feelings. Task-oriented training is aimed at improving the control strategy by solving difficulties through various measures.

In general, a variety of techniques, including Bobath approach, Roods approach, Proprioceptive neuromuscular facilitation techniques, motor relearning program, functional approaches, stretching exercises, therapeutic massage, constrain induced movement therapy, range of motion exercises, myofascial release, and strengthening exercises have been in practice for recovery of the affected limb functional mobility in patients with stroke. This study will evaluate the effects of music therapy along with task oriented training on balance and functional independence in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

Age 40-60 years Both males and females Diagnosed stroke patients Chronic stage (after 6 months of onset) Individuals with Burg Balance Score ≥ 20 ≤ 40 Functional Independence Measure score up to 3 (moderate assistance) Able to understand command Mini mental status examination score of over 20

Exclusion Criteria:

Systematic Disorder e.g. Rheumatoid arthritis Unstable Angina Coexisting physical impairments e.g. limb amputation Any previous history of neurological disease other than stroke e.g. Parkinson's Any previous history of fractures Hearing or perception deficits

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Balance | Change in Balance score will be measured at baseline, at 4th week, at 8th week
  Dynamic and static balance will be measured by Berg Balance Scale
Functional Independence | Change in functional independence will be measured at baseline, at 4th week, at 8th week
  Functional Independence will be measured by Functional Independence Measure

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Ahmad, PhD, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Immediately after publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending on 36th month